CLINICAL TRIAL: NCT03447379
Title: Short-term Dual Antiplatelet Therapy After Deployment of Bioabsorbable Polymer Everolimus-eluting Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Bumkee Hong, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-2017-0230
Record Dates: First submitted 2017-12-01; First posted 2018-02-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2022-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- P2Y12 antagonist monotherapy (Experimental): P2Y12 antagonist monotherapy after 3-month DAPT
  Interventions: Drug: P2Y12 antagonist monotherapy
- Aspirin + P2Y12 antagonist (Active Comparator): Aspirin + P2Y12 antagonist after 3-month DAPT
  Interventions: Drug: Aspirin plus P2Y12 antagonist

INTERVENTIONS:
Drug: P2Y12 antagonist monotherapy — P2Y12 inhibitor(Clopidogrel 75mg/day or Ticagrelor 180mg/day) for 9months after 3 months of DAPT(Aspirin 100mg/day + Clopidogrel 75mg/day or Aspirin 100mg/day + Ticagrelor 180mg/day)
  Arms: P2Y12 antagonist monotherapy
Drug: Aspirin plus P2Y12 antagonist — DAPT(Aspirin 100mg/day + Clopidogrel 75mg/day or Aspirin 100mg/day + Ticagrelor 180mg/day) for a year
  Arms: Aspirin + P2Y12 antagonist

SUMMARY:
To compare the clinical outcomes of P2Y12 antagonist monotherapy with aspirin plus P2Y12 antagonist following 3-month of DAPT in patients undergoing PCI with bioabsorbable polymer Everolimus-eluting stents (Synergy®)

ELIGIBILITY:
Inclusion Criteria:

1. Age 19+
2. Patients treated with a new generation of Evelorimus-eluting stents (Synergy®)
3. Patients who understand the content of the subject description and voluntarily sign the subject

Exclusion Criteria:

1. Age 86+
2. Hemodynamically unstable patient
3. Severe hypersensitivity reactions to aspirin, clopidogrel, ticagrelor, everolimus, contrast agent
4. Patients at high risk of bleeding, anemia, thrombocytopenia
5. Patients requiring oral anticoagulants
6. Pregnant women or women of childbearing age
7. Life expectancy is less than one year
8. Patients receiving a potent CYP3A4 inhibitor (eg, ketoconazole, clarithromycin, napjodone, ritonavir, atazanavir)
9. Patients with a history of intracranial hemorrhage
10. Patients with moderate to severe hepatic impairment
11. Patients underwent coronary intervention with stenting within 1 year
12. Patients with left-main lesions requiring coronary intervention
13. Patients with chronic stricture lesions requiring treatment
14. Patients with in-stent restenosis in a lesion requiring treatment
15. Patients with bifurcation lesions requiring stenting in lateral branches
16. Patients with lesions requiring more than 3 stents

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1452 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular clinical events (MACCE) | between 3 and 12 month after the procedure
  cardiovascular-related death, myocardial infarction, stent thrombosis, stroke, or target lesion revascularization
Major bleeding | between 3 and 12 month after the procedure
  The Bleeding Academic Research Consortium (BARC) type 3 or 5

CONTACTS AND LOCATIONS:
Overall Officials: Bumkee Hong, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, Souel, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Min PK, Kang TS, Cho YH, Cheong SS, Kim BK, Kwon SW, Park WJ, Lee JH, Kim W, Lee WS, Yoon YW, Lee BK, Kwon HM, Hong BK; SHARE Investigators. P2Y12 Inhibitor Monotherapy vs Dual Antiplatelet Therapy After Deployment of a Drug-Eluting Stent: The SHARE Randomized Clinical Trial. JAMA Netw Open. 2024 Mar 4;7(3):e240877. doi: 10.1001/jamanetworkopen.2024.0877. PMID 38451525